CLINICAL TRIAL: NCT06987344
Title: Field-based Closed Kinetic Chain Training With Progressive Eccentric Time Under Tension: Effects on Knee Strength and Lower Limb Viscoelasticity in Soccer Players: a Randomized Controlled Trial
Brief Title: How Eccentric Closed Chain Training Affects Knee Strength and Muscle Properties in Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Americas (Other)
Responsible Party: Principal Investigator, Maximiliano Torres-Banduc, Principal Investigator, University of Americas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2025015
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: Exercise therapy; Muscle strength; Lower extremity; Tendons

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Control Group (Active Comparator): Maintained their customary daily activities and regular soccer training routines: Trained three times a week, two days were dedicated to functional and tactical on-field training, while the third day was reserved for a two-hour gym session focused on flexibility, muscular strength, and endurance development.
  Interventions: Other: Regular soccer training routines
- Closed Kinetic Chain Group (Experimental): In addition to the same activities as the active cotrol group, participants performed five to seven different closed kinetic chain drills during the two days of field-based training, completing two to three sets per drill and eight to fourteen repetitions per set. The training volume underwent gradual increments over the course of every week. The total training volume for externally loaded CKC exercises was calculated by summing sets × repetitions × load (kg), yielding a cumulative volume of approximately 10,863 kg over 12 sessions. For exercises involving bodyweight or elastic resistance, training volume was estimated using time under tension (TUT), computed as the product of repetitions and eccentric phase duration. The cumulative TUT throughout the 6-week protocol amounted to 9,300 seconds (155 minutes) of eccentric loading.
  Interventions: Other: Field-based closed kinetic chain exercise with progressively increased time under tension; Other: Regular soccer training routines

INTERVENTIONS:
Other: Field-based closed kinetic chain exercise with progressively increased time under tension — This intervention is uniquely characterized by the integration of field-based closed kinetic chain (CKC) exercises with a systematically increased eccentric time under tension (TUT), specifically tailored for university-level soccer players. Unlike conventional strength training protocols, which are often gym-based and rely on traditional resistance machines or free weights, this program emphasizes functional, sport-specific movement patterns performed on the field, enhancing ecological validity and transfer to soccer performance.
  Arms: Closed Kinetic Chain Group
Other: Regular soccer training routines — Trained three times a week: two days were dedicated to functional and tactical on-field training, while the third day was reserved for a two-hour gym session focused on flexibility, muscular strength, and endurance development.

SUMMARY:
The goal of this study is to learn whether a 6-week lower-body training program using closed kinetic chain (CKC) exercises with slow, controlled movements (called "eccentric time under tension") can improve leg muscle strength and muscle-tendon viscoelastic properties in male university soccer players.

The Main Questions Are:

1. Does this type of training improve knee strength?
2. Does it change the way muscles and tendons respond to movement or pressure?

What Will Participants Do?

1. Join one of two groups: one does the CKC training program, the other continues regular soccer training
2. Train twice a week for 6 weeks
3. Have their leg strength tested using special equipment
4. Have their muscle and tendon properties measured with a handheld device

DETAILED DESCRIPTION:
This randomized controlled trial investigated the effects of a 6-week, field-based closed kinetic chain (CKC) exercise program with progressively increased eccentric time under tension (TUT) on isokinetic knee performance and lower limb muscle-tendon viscoelastic properties in male university soccer players.

A total of 24 healthy participants were randomly assigned (1:1) to either an intervention group performing supervised CKC exercises or an active control group that maintained routine soccer training. The CKC training was performed twice per week and included progressive increases in eccentric phase duration and external loading. Training volume was quantified using both mechanical load and eccentric TUT. Each session lasted approximately 35 minutes and included a variety of multi-joint, bilateral and unilateral exercises performed on a soccer field.

Baseline and post-intervention assessments were conducted using:

Isokinetic dynamometry (Biodex System 3 Pro) to measure concentric peak torque, mean power, and agonist/antagonist ratio at 60°/s.

MyotonPRO handheld myotonometer to assess oscillation frequency and stiffness of specific lower limb muscles (VM, VL, ST, GM) and tendons (Achilles, patellar).

Muscle and tendon assessments were performed following standardized anatomical landmarks. To ensure data reliability, repeated trials were used and measurements with high variability were repeated. Pre-testing familiarization was implemented to reduce learning effects.

The statistical approach included a two-way repeated measures ANOVA to compare group (CKC vs. control) and time (pre vs. post) effects. Holm-Sidak post hoc tests were applied when appropriate, and effect sizes were interpreted using eta squared (η²). All data analyses were conducted using JASP software (v0.18.3).

The protocol was reviewed and approved by an institutional ethics committee , and written informed consent was obtained from all participants. No serious adverse events were reported, and dropout was minimal (n = 4). No dietary interventions were applied; however, participants were instructed to maintain consistent routines throughout.

ELIGIBILITY:
Inclusion Criteria:

* Absence of any medical conditions that could compromise their ability to participate.
* Active membership in their university's soccer team for a minimum of one year.

Exclusion Criteria:

* Musculoskeletal injuries reported in the two months prior to the start of the study.
* Surgical interventions involving the lower limbs within the past year.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the rotational peak torque relative to body mass at 6 weeks | From enrollment to the end of closed kinetic chain training protocol at 6 weeks
  Assessed using a Biodex® System 3 Pro isokinetic dynamometer (Shirley, NY, USA), with a validated accuracy of ±1%.
  Testing was performed at 60°/s angular velocity, a standard velocity for evaluating maximal voluntary muscle contraction.
  Participants were seated with their hips and knees at approximately 90° flexion. The dominant leg was tested and stabilized using straps at the trunk, thigh, and lower leg. Gravity correction was applied prior to testing.
  Following a 5-minute warm-up and 3 submaximal practice repetitions, each participant performed 3 maximal concentric repetitions of knee extension and flexion.
  The dominant leg was defined as the preferred leg for kicking, confirmed via observation of a standardized ball-kicking task.
Change from baseline in the rotational mean power at 6 weeks | From enrollment to the end of closed kinetic chain training protocol at 6 weeks
  Assessed using a Biodex® System 3 Pro isokinetic dynamometer (Shirley, NY, USA), with a validated accuracy of ±1%.
  Testing was performed at 60°/s angular velocity, a standard velocity for evaluating maximal voluntary muscle contraction.
  Participants were seated with their hips and knees at approximately 90° flexion. The dominant leg was tested and stabilized using straps at the trunk, thigh, and lower leg. Gravity correction was applied prior to testing.
  Following a 5-minute warm-up and 3 submaximal practice repetitions, each participant performed 3 maximal concentric repetitions of knee extension and flexion.
  The dominant leg was defined as the preferred leg for kicking, confirmed via observation of a standardized ball-kicking task.

SECONDARY OUTCOMES:
Change from baseline in the agonist/antagonist strength ratio at 6 weeks | From enrollment to the end of closed kinetic chain training protocol at 6 weeks
  Assessed using a Biodex® System 3 Pro isokinetic dynamometer (Shirley, NY, USA), with a validated accuracy of ±1%. Was calculated as the percentage of knee flexor peak torque relative to knee extensor peak torque.
  Testing was performed at 60°/s angular velocity, a standard velocity for evaluating maximal voluntary muscle contraction.
  Participants were seated with their hips and knees at approximately 90° flexion. The dominant leg was tested and stabilized using straps at the trunk, thigh, and lower leg. Gravity correction was applied prior to testing.
  Following a 5-minute warm-up and 3 submaximal practice repetitions, each participant performed 3 maximal concentric repetitions of knee extension and flexion.
  The dominant leg was defined as the preferred leg for kicking, confirmed via observation of a standardized ball-kicking task.
Change from Baseline in the muscle oscillation frequency at 6 weeks | From enrollment to the end of closed kinetic chain training protocol at 6 weeks
  Evaluated using the MyotonPRO® handheld myotonometer (Myoton AS, Estonia), a non-invasive digital palpation device validated for muscle and tendon assessment.
  Muscles assessed on the dominant leg included:
  Muscles: Vastus Medialis (VM), Vastus Lateralis (VL), Semitendinosus (ST), Gastrocnemius Medialis (GM)
  Participants were positioned supine or prone, depending on the target tissue. The device probe was applied perpendicularly to the skin over the anatomical landmark recommended by the manufacturer.
  Each site was measured three times, and the mean value was used for analysis. Measurements were repeated if the coefficient of variation exceeded 10%.
Change from Baseline in the stiffness at 6 weeks | From enrollment to the end of closed kinetic chain training protocol at 6 weeks
  Evaluated using the MyotonPRO® handheld myotonometer (Myoton AS, Estonia), a non-invasive digital palpation device validated for muscle and tendon assessment.
  Muscles and tendons assessed on the dominant leg included:
  Muscles: Vastus Medialis (VM), Vastus Lateralis (VL), Semitendinosus (ST), Gastrocnemius Medialis (GM) Tendons: Patellar Tendon (PT), Achilles Tendon (AT)
  Participants were positioned supine or prone, depending on the target tissue. The device probe was applied perpendicularly to the skin over the anatomical landmark recommended by the manufacturer.
  Each site was measured three times, and the mean value was used for analysis. Measurements were repeated if the coefficient of variation exceeded 10%.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Movement Analysis Laboratory, Viña del Mar, V región/Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: No
Will be reported or made available upon reasonable request.